CLINICAL TRIAL: NCT00139906
Title: A Randomized, Double-Blind, Placebo-Controlled, Twice Daily Titration Study of the Safety and Tolerability of Bifeprunox in Subjects With Schizophrenia
Brief Title: Twice Daily Titration Study of Bifeprunox in Subjects With Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Solvay Pharmaceuticals (Industry)
Collaborators: H. Lundbeck A/S (Industry); Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: S154.2.016
Record Dates: First submitted 2005-08-30; First posted 2005-08-31 (Estimated); Last update posted 2015-01-16 (Estimated); Status verified 2006-03

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Titration Study; Schizophrenia; BID dosing; Pharmacokinetic
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — bifeprunox

INTERVENTIONS:
Drug: Bifeprunox

SUMMARY:
This study is to assess the safety and tolerability of a five-day titration schedule (using twice daily dosing for the first three days) to achieve the highest proposed dose of 40 mg daily. The study duration is two months.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have current diagnosis of Schizophrenia or Schizoaffective disorder
* Body weight of 100-250 lbs
* Male or females
* 18-55 years of age

Exclusion Criteria:

* Subjects who are acutely psychotic
* Subjects with current Axis I primary psychiatric diagnosis other than schizophrenia, at significant risk of suicide

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 2005-08; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Director Solvay, Study Director — Solvay Pharmaceuticals
Locations (1):
- Site 1, National City, California, United States